CLINICAL TRIAL: NCT05697146
Title: Ribociclib Real-world Treatment Patterns and Clinical Outcomes Among Women With HR+/HER2- Advanced or Metastatic Breast Cancer in France: a National, Multicenter, Prospective, Non-interventional Study
Brief Title: Ribociclib Real-world Treatment Patterns and Clinical Outcomes Among Women With HR+/HER2- Advanced or Metastatic Breast Cancer in France
Acronym: RosaLEE
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011AFR01
Record Dates: First submitted 2022-11-08; First posted 2023-01-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: HR+/HER2- advanced or metastatic breast cancer; RosaLEE; NIS; France; Ribociclib
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- ribociclib + ET: Women prescribed ribociclib + Endocrine Therapy (ET)
  Interventions: Other: ribociclib + ET

INTERVENTIONS:
Other: ribociclib + ET — There is no treatment allocation. Patients administered ribociclib + endocrine Therapy (ET) by prescription will be enrolled.

SUMMARY:
This study is a national, multicenter, prospective, non-interventional study in women with HR+/HER2- locally advanced or metastatic breast cancer (BC), for which a prior clinical decision to initiate ribociclib + endocrine therapy (ET) treatment according to the marketing authorization has been taken and was taken independent and prior to study participation decision.

DETAILED DESCRIPTION:
Included patients will be followed until the end of study, death or lost to follow-up even if ribociclib and ET are discontinued. The end of the study is defined as 3 years after the first visit of the last patient included (Last Patient First Visit [LPFV]). The total duration of the study will be 4 years and half (18 months of inclusion + 3 years of follow-up). Thus, a patient included at the beginning of the inclusion period will be followed for 4 years and half and a patient included at the end of the inclusion period will be followed for at least 3 years.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria will be included in the RosaLEE study:

1. Adult women aged ≥ 18 years old at inclusion.
2. Pre-/Peri-/Postmenopausal women with locally advanced or metastatic HR+/HER2- BC.
3. Prior clinical decision (independent of study participation)to initiate ribociclib + ET treatment according to the marketing authorization.
4. Patients having given their non-objection to participate in the study.
5. Patients presenting with medical conditions to be treated with ribociclib + ET according to the summary of product characteristics.

Exclusion Criteria:

1. Patients for whom ribociclib + AI in treatment combination has been initiated before inclusion.
2. Patients for whom ribociclib + fulvestrant in treatment combination has been initiated before inclusion.
3. Patients for whom AI or fulvestrant in monotherapy has been initiated > 28 days before inclusion.
4. Participation in any clinical study involving investigational therapy except for the Trans-RosaLEE study, conducted by the IPC.
5. Patient who is pregnant or has expressed desire for pregnancy during Ribociclib treatment.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pre-/perimenopausal and postmenopausal women with HR+/HER2- advanced or metastatic breast cancer
Study Population: Advanced HR+/HER2- breast cancer population treated with ribociclib in France
Sampling Method: Non-Probability Sample
Enrollment: 1018 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients by initial dose of ribociclib | Baseline
  Proportion of patients by initial dose of ribociclib to be collected
Proportion of patients by endocrine therapy partner | Baseline, up to 54 months
  Proportion of patients by endocrine therapy partner to be collected(e.g., tamoxifen, letrozole, fulvestrant, anastrozole, exemestane, LHRH agonist)
Proportion of patients for each line of treatment with ribociclib | Baseline
  Proportion of patients for each line of treatment with ribociclib (1L, 2L, >2L) to be collected

SECONDARY OUTCOMES:
Progression Free Survival (PFS) by treatment line and endocrine partner | month 12, month 24, month 36, up to 54 months
  Progression free survival (PFS): time from the date of treatment initiation with ribociclib to the date of the first documented disease progression or death due to any cause, whichever occurs first; if a patient has not had an event, the PFS will be censored at the date of the last adequate tumor assessment (RECIST 1.1).
Overall Survival (OS) | month 12, month 24, month 36, up to 54 months
  Overall survival: time from the date of treatment initiation with ribociclib until death due to any cause; if a patient is not known to have died, then the OS will be censored at the latest date the patient was known to be alive.
Identify prognostic factors influencing the OS and PFS | Up to 54 months
  Prognostic factors influencing the OS and PFS will be listed
Proportion of patients with adjuvant treatment and type of treatment | Up to 54 months
  Proportion of patients with adjuvant treatment and type of treatment to be collected
Proportion of patients treated with chemotherapy/ET/targeted therapy and type of local treatment | Up to 54 months
  Proportion of patients treated with chemotherapy/ET/targeted therapy and type of local treatment to be collected
Proportion of patients by menopausal status | Up to 54 months
  Proportion of patients by menopausal status (pre-/perimenopausal patients versus postmenopausal patients)
Proportion of de novo metastatic patients, 1L, 2L and >2L at ribociclib initiation | Up to 54 months
  Proportion of de novo metastatic patients, 1L, 2L and >2L at ribociclib initiation to be collected
Proportion of patients with complete response (CR)/partial response (PR)/stable disease (SD)/progressive disease (PD)/unknown | Up to 54 months
  Proportion of patients with complete response (CR)/partial response (PR)/stable disease (SD)/progressive disease (PD)/unknown to be collected
Overall response rate | Up to 54 months
  Overall response rate, defined as the proportion of patients with best overall response or complete response (CR) or partial response (PR) according to RECIST 1.1.
In the subgroup of patients with visceral metastasis: median PFS | Up to 54 months
  Progression free survival (PFS): time from the date of treatment initiation with ribociclib to the date of the first documented disease progression or death due to any cause, whichever occurs first; if a patient has not had an event, the PFS will be censored at the date of the last adequate tumor assessment (RECIST 1.1).
In the subgroup of patients with visceral metastasis: PFS rate | Up to 54 months
  Progression free survival (PFS): time from the date of treatment initiation with ribociclib to the date of the first documented disease progression or death due to any cause, whichever occurs first; if a patient has not had an event, the PFS will be censored at the date of the last adequate tumor assessment (RECIST 1.1).
In the subgroup of patients with visceral metastasis: median OS | Up to 54 months
  Overall survival: time from the date of treatment initiation with ribociclib until death due to any cause; if a patient is not known to have died, then the OS will be censored at the latest date the patient was known to be alive.
In the subgroup of patients with visceral metastasis: OS rate | Up to 54 months
  Overall survival: time from the date of treatment initiation with ribociclib until death due to any cause; if a patient is not known to have died, then the OS will be censored at the latest date the patient was known to be alive.
In the subgroup of patients with visceral metastasis: proportion of patients with CR/PR/SD/PD/unknown | Up to 54 months
  In the subgroup of patients with visceral metastasis: proportion of patients with complete response (CR)/partial response (PR)/stable disease (SD)/progressive disease (PD)/unknown to be collected
Sequential PFS (S-PFS) | month 12, month 24, month 36, up to 54 months
  Sequential progression free survival: time from the date of treatment initiation with ribociclib to the date of the second and subsequent documented progression or death due to any cause, whichever occurs first.
Time to chemotherapy since ribociclib initiation | Up to 54 months
  Time to chemotherapy since ribociclib initiation to be collected
Proportion of patients with ribociclib dose adjustment after treatment initiation and reason(s) | Up to 54 months
  Proportion of patients with ribociclib dose adjustment after treatment initiation; adjustment type (dose modifications/interruptions during treatment) and reason(s) for dose modifications/interruptions).
Treatment exposure to ribociclib | Up to 54 months
  Treatment exposure to ribociclib: time from treatment initiation to treatment discontinuation.
Reason(s) for discontinuation | Up to 54 months
  Treatment discontinuation: permanent cessation of the treatment received, for any reason.
In the subgroup of oligometastatic patients at inclusion: proportion of patients treated with local treatment | Up to 54 months
  In the subgroup of oligometastatic patients at inclusion: proportion of patients treated with local treatment and treatment outcome to be collected
Proportion of visits in the site versus proportion of remote visits | Up to 54 months
  Proportion of visits in the site versus proportion of remote visits to be collected
Proportion of patients with at least one hospitalization | Up to 54 months
  Proportion of patients with at least one hospitalization to be collected
EuroQol 5-Dimension Questionnaire5-level version (EQ-5D-5L) scores | Up to 54 months
  EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3=moderate problems, 4= severe problems, and 5= extreme problems. Higher scores indicated greater levels of problems across each of the five dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (71):
- France (71):
  - Novartis Investigative Site, Nice, Alpes Maritimes
  - Novartis Investigative Site, Marseille, Bouches Du Rhone
  - Novartis Investigative Site, Dijon, Cote D Or
  - Novartis Investigative Site, Saint-Denis, France
  - Novartis Investigative Site, Valenciennes, France
  - Novartis Investigative Site, Saint-Cloud, Hauts De Seine
  - Novartis Investigative Site, Grenoble, Isere
  - Novartis Investigative Site, Reims, Marne
  - Novartis Investigative Site, Toulon, Val De Marne
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Argenteuil
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Bayonne
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Béziers
  - Novartis Investigative Site, Brive-la-Gaillarde
  - Novartis Investigative Site, Cannes
  - Novartis Investigative Site, Carcassonne
  - Novartis Investigative Site, Chalon-sur-Saône
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Champigny-sur-Marne
  - Novartis Investigative Site, Cherbourg
  - Novartis Investigative Site, Cholet
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Colmar
  - Novartis Investigative Site, Compiègne
  - Novartis Investigative Site, Corbeil-Essonnes
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Dechy
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Dunkirk
  - Novartis Investigative Site, Eaubonne
  - Novartis Investigative Site, Fréjus
  - Novartis Investigative Site, Gleizé
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, Libourne
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Lyon 08
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Metz
  - Novartis Investigative Site, Metz-Tessy
  - Novartis Investigative Site, Montbelliard
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nancy
  - Novartis Investigative Site, Neuilly-sur-Seine
  - Novartis Investigative Site, Niort
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Osny
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Perpignan
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Dizier
  - Novartis Investigative Site, Saint-Etienne
  - Novartis Investigative Site, Saint-Nazaire
  - Novartis Investigative Site, Saint-Pierre
  - Novartis Investigative Site, Saint-Vallier
  - Novartis Investigative Site, Sarcelles
  - Novartis Investigative Site, Soyaux
  - Novartis Investigative Site, St-Malo
  - Novartis Investigative Site, Suresnes
  - Novartis Investigative Site, Thionville
  - Novartis Investigative Site, Toulon La Seyne
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Valence
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
  - Novartis Investigative Site, Vantoux
  - Novartis Investigative Site, Villejuif
  - Novartis Investigative Site, Villeurbanne